CLINICAL TRIAL: NCT04289155
Title: Individual Patient Compassionate Use of GX-I7
Status: No longer available | Type: Expanded Access
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GX-I7_TP
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Glioblastoma; High Grade Glioma; Recurrent Glioblastoma; Melanoma; Advanced Cancer
MeSH Terms: conditions — Glioblastoma; Glioma; Melanoma | interventions — efineptakin alfa

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: GX-I7 — patients will receive the assigned dose of GX-I7 intramuscular injection every 4~12 weeks

SUMMARY:
Compassionate use of GX-I7 for patients with serious life-threatening illness that have exhausted all available therapies, with no other therapy options.

DETAILED DESCRIPTION:
This program is being offered on a patient by patient basis and will require company, Institutional Review Board/Independent Ethics Committee and Single Patient IND approval.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Kangnam St. Mary's Hospital, Seoul, South Korea